CLINICAL TRIAL: NCT07004192
Title: The Role of hCG in Thawed Embryo Transfer
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fertility Center of Las Vegas (Industry)
Responsible Party: Principal Investigator, Bruce Shapiro M.D., Medical Director, Fertility Center of Las Vegas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FCLV 2025-1
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Infertility (IVF Patients)
Keywords: Thawed embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- hCG Group (Experimental): This group receives one injection of hCG.
  Interventions: Drug: HCG injection
- No hCG Group (Active Comparator): This arm receives no hCG.
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: HCG injection — 5000 IU hCG injection
  Arms: hCG Group
Other: No intervention — No hCG administered in this group.
  Arms: No hCG Group

SUMMARY:
This prospective randomized trial will assess the relevance, if any, of a corpus luteum induced by hCG in transfers of thawed embryos.

DETAILED DESCRIPTION:
The current study is designed to carefully isolate the effect of a corpus luteum by ensuring that the presence or absence of a corpus luteum is the only difference between two study arms. This should be reliably achieved by administering an injection of hCG in one study arm, while the other study arm has identical treatment except for omitting the hCG.

ELIGIBILITY:
Inclusion Criteria:

1. Female adult expecting to receive transfer of a thawed embryo.
2. At least one available frozen blastocyst of transferrable quality.
3. Non-menopausal female with at least one antral follicle.
4. Use of pre-implantation genetic testing (PGT), embryos derived from donor oocytes and/or donor sperm, a gestational carrier, and history of prior transfer(s) regardless of outcome are allowed.
5. Subsequent embryo transfers after failed transfers under this study are allowed, but not after a transfer that has resulted in ongoing pregnancy at ten weeks gestation under this study.

Exclusion Criteria:

1. Minors (age<18 years).
2. Use of embryo(s) frozen at another center.
3. Patient insistent on transfer of two embryos.
4. Patient or partner unable to provide informed consent in English.
5. Patient already enrolled in any other research study for her embryo transfer.
6. History of anti-phospholipid syndrome or any other indication for use of Lovenox in pregnancy.
7. Patient for whom the physician assesses this protocol is inappropriate or unsafe.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Third trimester of pregnancy
  Mean arterial pressure measured in third trimester of pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Center of Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to do so in approved protocol.